CLINICAL TRIAL: NCT02933034
Title: Clinical Trial of Manganese-Enhanced MRI (MEMRI) to Assess Peri-Infarct Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Phillip C. Yang, MD, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 28508
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: ISCHEMIC CARDIOMYOPATHY
Keywords: ISCHEMIC OR CORONARY HEART DISEASE; MYOCARDIAL INFARCTION; MAGNETIC RESONANCE IMAGING; DELAYED GADOLINIUM ENHANCEMENT MRI; MANGANESE-ENHANCED MRI; INFARCT VOLUME/SIZE; ALL CAUSE MORTALITY; VENTRICULAR ARRHYTHMIAS
MeSH Terms: conditions — Myocardial Infarction | interventions — EVP 1001-1; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Coronary Disease (Experimental): Participant receive 2 cardiac MRI procedures: MEMRI and DEMRI.
  Interventions: Drug: Manganese-enhanced MRI contrast reagent; Drug: Gadolinium-enhanced MRI contrast reagent

INTERVENTIONS:
Drug: Manganese-enhanced MRI contrast reagent — MRI using manganese-enhanced MRI contrast reagent (manganese 0.28 mL/kg).
  Other Names: EVP 1001-1
Drug: Gadolinium-enhanced MRI contrast reagent — MRI using gadolinium-enhanced MRI contrast reagent (gadolinium 0.2 mmol/kg).
  Other Names: GD-DTPA

SUMMARY:
The purpose of this study is to evaluate the safety and tolerance of a new intravenous diagnostic agent, SeeMore or EVP 1001-1, in patients with Cardiovascular Disease (MEMRI scan). The initial phase of this study, NCT01989195 enrolling a total of 6 patients, has been closed. This second phase adds 10 patients in a safety cohort and 60 additional patients for a total of 70 patients.

DETAILED DESCRIPTION:
This is an open-label, baseline-controlled study to be conducted. Adult male or nonpregnant female patients who have been referred for evaluation of dilated cardiomyopathy, ischemic cardiomyopathy, non-ischemic cardiomyopathy, atrial arrhythmia and also patients who have received stem cell therapy related to both ischemic and dilated cardiomyopathy (under different trials) will be recruited. An initial cohort study of 6 patients to conduct safety evaluation was conducted before proceeding with 60 additional patients. In the initial cohort, a patient was dosed based on the Phase 1 and 2 clinical trial data evaluation completed by Eagle Vision Pharmaceutical, Inc. Subjects were excluded if they had received an investigational device within 30 days prior to administration of EVP1001-1; had a history of drug abuse or alcoholism; were taking a digitalis preparation; had a history of torsades; had New York Heart Association (NYHA) Grade IV heart failure; had abnormal liver function tests or a history of liver disease; had uncontrolled hypertension; had abnormal calcium, potassium or hemoglobin values at baseline; if they develop a cardiac arrhythmia prior to or during either of the exercise tests-- EVP1001-1 was not administered. The same parameters will apply to the new group of subjects.

Prior to entry into this study, all subjects will sign an Informed Consent and will undergo a physical examination including medical history, details regarding their cardiac history, prescription and over-the-counter drug questionnaire, vital signs, electrocardiogram (ECG), evaluation of the major organ systems, hematology, serum chemistries, and urinalysis. In addition, female subjects will undergo a serum pregnancy test.

Starting 30 minutes before the cardiac MRI scan (CMR), the subjects will take a 16 mg tablet of ondansetron by mouth. CMR imaging will subsequently take place and then EVP1001-1 will then be administered approximately 15 minutes into the scan for contrast enhanced images. EVP1001-1 will be administered intravenously over approximately one minute. The subjects will each receive 0.28 mL/kg of EVP 1001-1. All subjects will be monitored closely from before ondansetron administration until their discharge from the imaging center. Following MEMRI, delayed-enhanced MRI (DEMRI scan) is performed using 0.2 mmol/kg.

We will compare the two different contrast enhanced images (EVP1001-1 vs gadolinium (GD)) in determining the non-viable (infarct core), peri-infarct, and total infarct size of myocardial tissue.

ELIGIBILITY:
Inclusion Criteria:

All subjects to be entered must:

* be at least 18 years of age.
* if female, be nonpregnant as evidenced by a serum pregnancy test and using a medically-approved method of birth control, or post-menopausal or surgically sterile
* provide written informed consent after having received oral and written information about the study
* be in stable health based on medical history, examination and tests

Exclusion Criteria:

have a positive pregnancy test (females)

* received an investigational drug or device within 30 days prior to administration of SeeMore
* have known hypersensitivity to ondansetron or other selective serotonin 5HT3 receptor blockers
* have a history of drug abuse or alcoholism
* are taking a digitalis preparation or calcium channel blocker
* have a history of torsades or prolonged QT/QTc interval
* have NYHA Grade IV heart failure
* have abnormal liver function tests or a history of liver disease
* have uncontrolled hypertension (Systolic Blood Pressure > 140 or Diastolic BP > 90 consistently at baseline)
* have abnormal baseline potassium or calcium values or hemoglobin less than 10 g/dl
* are noncompliant or otherwise unlikely to perform as required by the protocol
* have pretest likelihood of CAD for which the requisite number of subjects have been entered
* develop an arrhythmia prior to or during either of the exercise tests; SeeMore should not be administered.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip C Yang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Coronary Disease Patients: Participants receive 2 cardiac MRI procedures: manganese-enhanced MRI (MEMRI; manganese 0.28 mL/kg as reagent); and delayed-enhanced MRI (DEMRI; gadolinium 0.2 mmol/kg as reagent).
Period: Overall Study
Arm/Group | Coronary Disease Patients
Started | 33
Received Both MEMRI and DEMRI Scans | 24
Completed | 24
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Participants who had both MEMRI and DEMRI scans were considered evaluable for baseline characteristics
Groups:
- Coronary Disease Patients: Participants receive 2 cardiac MRI procedures: MEMRI (manganese 0.28 mL/kg as reagent); and DEMRI (gadolinium 0.2 mmol/kg as reagent).
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11
  Asian | 4
  South Asian | 6
  Latino | 3
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Infarct Size of MEMRI Versus DEMRI Scans
Description: MEMRI is an assessment of non-viable myocardial tissue and evaluates core infarct size. DEMRI is an assessment of fibrotic tissue and evaluates the total infarct size. The difference between these two measurements evaluates the size of peri-infarct region consisting of mixed components of injured but viable cardiomyocytes and fibrosis.
Time Frame: Day of MEMRI and DEMRI scans (up to 3 hours per scan, performed on the same day or up to 7 days apart)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: percentage of left ventricle
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
percentage of left ventricle
  MEMRI | 12.2 (7.3)
  DEMRI | 18.9 (11.9)
Statistical Analysis 1: Comparison: Coronary Disease Patients; Comparison of infarct size using MEMRI versus DEMRI scan; Test type: Other; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure during MEMRI scan as a measure of manganese contrast reagent safety. Normal reference range: 90-120 mmHg.
Time Frame: Before, during, and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
mmHg
  Baseline | 121.8 (16.4)
  During MRI | 160.9 (24.4)
  Post MRI | 124.4 (18.3)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure during MEMRI scan as a measure of manganese contrast reagent safety. Normal reference range: 60-80 mmHg.
Time Frame: Before,during, and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
mmHg
  Baseline | 71.8 (9.1)
  During MRI | 92.6 (10.8)
  Post MRI | 66.2 (10.0)

4. Secondary Outcome: Heart Rate
Description: Heart rate during MEMRI scan as a measure of manganese contrast reagent safety. Normal reference range: 60 and 100 beats per minute.
Time Frame: Before,during, and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
beats per minute
  Baseline | 66.3 (9.9)
  During MRI | 82.8 (15.1)
  Post MRI | 66.2 (10.0)

5. Secondary Outcome: QT Interval
Description: QT interval during MEMRI scan as a measure of manganese contrast reagent safety. QT is a measurement of heart function that is dependent on heart rate, so QTc is mainly used for diagnosis rather than QT. Normal reference range was considered to be 360-450 milliseconds for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
milliseconds
  Baseline | 414.7 (40.1)
  Post MRI | 412.6 (38.2)

6. Secondary Outcome: Corrected QT (QTc)
Description: Corrected QT (QTc) interval during MEMRI scan as a measure of manganese contrast reagent safety. QTc is a measurement of heart function and is mainly used for diagnosis rather than QT, because QT is dependent on heart rate. Normal reference range was considered to be 360-450 milliseconds for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
milliseconds
  Baseline | 435.7 (34.5)
  Post MRI | 440.5 (37.3)

7. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: ALT levels during MEMRI scan as a measure of manganese contrast reagent safety. ALT is a measurement of liver function. Normal reference range was considered to be <60 U/L for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
U/L
  Baseline | 37.8 (18.4)
  Post MRI | 35.1 (12.6)

8. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: AST levels during MEMRI scan as a measure of manganese contrast reagent safety. AST is a measurement of liver function. Normal reference range was considered to be <40 U/L for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
U/L
  Baseline | 26.1 (12.4)
  Post MRI | 25.4 (9.1)

9. Secondary Outcome: Alkaline Phosphatase (ALP)
Description: ALP levels during MEMRI scan as a measure of manganese contrast reagent safety. ALP is a measurement of liver function. Normal reference range was considered to be <40-130 U/L for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
U/L
  Baseline | 80.8 (21.9)
  Post MRI | 79.8 (26.7)

10. Secondary Outcome: Total Bilirubin
Description: Total bilirubin levels during MEMRI scan as a measure of manganese contrast reagent safety. Total bilirubin is a measurement of liver function. Normal reference range was considered to be <1.4 mg/dL for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
mg/dL
  Baseline | 0.58 (0.21)
  Post MRI | 0.65 (0.30)

11. Secondary Outcome: Creatinine
Description: Creatinine levels during MEMRI scan as a measure of manganese contrast reagent safety. Creatinine is a measurement of kidney function. Normal reference range was considered to be 0.50-1.20 mg/dL for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
mg/dL
  Baseline | 1.04 (0.23)
  Post MRI | 1.10 (0.19)

12. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR levels during MEMRI scan as a measure of manganese contrast reagent safety. eGFR is a measurement of kidney function. Normal reference range was considered to be >60 ml/min/1.73m^2 for this study.
Time Frame: Before and after MEMRI scan (up to 3 hours)
Population: Participants who had both MEMRI and DEMRI scans are included in the analysis
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Coronary Disease Patients
Number analyzed (Participants) | 24
mL/min/1.73m^2
  Pre MRI | 75.4 (20.5)
  Post MRI | 70.5 (16.0)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (average 616 days)
Groups:
- Coronary Disease Patients: Participants receive 2 cardiac MRI procedures: MEMRI (manganese 0.28 mL/kg as a reagent); and DEMRI (gadolinium 0.2 mmol/kg as a reagent).
Arm/Group | Coronary Disease Patients
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 14/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coronary Disease Patients (N=33)
abdominal discomfort (Gastrointestinal disorders) | 1
abdominal pain (Gastrointestinal disorders) | 3
anxiety (Nervous system disorders) | 1
chest pain (General disorders) | 2
constipation (Gastrointestinal disorders) | 1
fatigue (General disorders) | 2
flushing (Vascular disorders) | 9
hypoglycemia (Metabolism and nutrition disorders) | 1
lip numbness (Nervous system disorders) | 1
malaise (General disorders) | 1
nausea (Gastrointestinal disorders) | 3
mild discomfort (General disorders) | 1
mild jaw pain (General disorders) | 1
mild weakness of feet (General disorders) | 1

LIMITATIONS AND CAVEATS:
The study did not meet its planned sample size of 70 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT02933034/Prot_SAP_000.pdf